CLINICAL TRIAL: NCT02926235
Title: Randomized Control Trial of Essential Amino Acid Supplementation in Protein Deficient Patients Following Total Knee Arthroplasty
Brief Title: Trial of Essential Amino Acid Supplementation in Protein Deficient Patients Following Total Knee Arthroplasty
Acronym: Amino Acid
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-067
Record Dates: First submitted 2016-06-24; First posted 2016-10-06 (Estimated); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Quad Atrophy
Keywords: Total Knee Arthroplasty
MeSH Terms: interventions — Amino Acids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amino Acid (Experimental): Patients will be asked to ingest 20g of EAA o two times a day between meals 1 week prior and 2 weeks postoperatively.
  Interventions: Drug: Amino Acid
- Placebo (Placebo Comparator): Patients will be asked to ingest 20g of placebo two times a day between meals 1 week prior and 2 weeks postoperatively.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Amino Acid — Treatment arm
  Arms: Amino Acid
Other: Placebo
  Arms: Placebo

SUMMARY:
The goal of this trial is to assess the efficacy of essential amino acids (EAA) on muscle atrophy and malnutrition compared to a placebo in patients following a total knee arthroplasty. The investigators specific objectives included analysis of (1) muscle strength, (2) change in malnutrition, (3) perioperative complications (4) physical activity.

DETAILED DESCRIPTION:
Three orthopedic surgeons will participate in the study (MBC, DJM, SAJ). The surgical procedure will be performed as per each surgeon's routine practice. Patients will be asked to ingest 20g of EAA or placebo two times a day between meals 1 week prior and 2 weeks postoperatively. Patients will be given a pill organizer that has two doses per day with either EAA or placebo. Thigh circumference will be measured at baseline, 2 weeks and 6 weeks post-operatively. The mid-thigh measurement will be taken while the patient stands erect with their feet slightly apart and their weight equally distributed. The girth measurement is taken perpendicular to the long axis of the thigh. The tape measure will be placed at the level midway between the trochanterion and tibiale laterale sites each time to ensure that the same location is measured each time. The investigators will measure strength using a handheld dynamometer and performing a straight leg raise and knee extension at 90 degrees on the operative and the non-operative leg preoperatively, 2 weeks and 6 weeks post-operatively. The medial and lateral epicondyles of the femur will be used to position the subject's knee joint through the axis of rotation on the dynamometer. Strength will be tested at 30, 45 and 60 degrees of flexion. Physical activity will be collected using the Knee Society Score at baseline and at 6 weeks postoperatively. After the trial is commenced, there will be no additional enrollment once study numbers have been met.

ELIGIBILITY:
Inclusion Criteria:

* All patients will be undergoing a primary unilateral total knee arthroplasty for a diagnosis of osteoarthritis

Exclusion Criteria:

* All patients who were wheelchair bound preoperatively
* All patients who cannot participate in an outpatient physical therapy program for 3 days per week after surgery

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-04; Primary Completion 2022-05-14 (Actual); Study Completion 2022-05-14 (Actual)

PRIMARY OUTCOMES:
Change Quad Strength | Change between preop and 6 weeks.
  As Measured by Quad circumference in inches

CONTACTS AND LOCATIONS:
Overall Officials: David Mayman, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States